CLINICAL TRIAL: NCT06026553
Title: A Randomized Blinded Placebo Controlled Trial Assessing Ketorolac (Toradol) at Oocyte Retrieval
Brief Title: Assessing Ketorolac (Toradol) at Oocyte Retrieval
Acronym: Alleviate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: TORA-IVF-01
Record Dates: First submitted 2023-08-22; First posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Infertility; Infertility, Female; Oocyte Retrieval; Postoperative Pain; Embryo Transfer
Keywords: Infertility, Female; In Vitro Fertilization; IVF; Oocyte Retrieval; Postoperative Pain Control; NSAID; Ketorolac; Non-Narcotic Analgesia
MeSH Terms: conditions — Infertility; Infertility, Female; Pain, Postoperative | interventions — Ketorolac; Ketorolac Tromethamine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Allocation group will not be disclosed to the patient or the physician or the nurse or the outcome assessor. The anesthesia provider administering the IV Ketorolac or Placebo will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard post-operative pain management + Ketorolac (Toradol) (Experimental): Subject will undergo an IVF cycle with ovarian hyperstimulation and oocyte retrieval. Standard protocols will be used for both study groups and involve administration of gonadotropins to stimulate ovarian follicle growth and regular monitoring with ultrasound and serum estradiol and progesterone levels until follicles reach a desired size. Human Chorionic Gonadotropin (HCG) or leuprolide acetate will be administered to trigger final oocyte maturation prior to oocyte retrieval under anesthesia. On the day of oocyte retrieval, the anesthesia provider will provide syringes of IV ketorolac (30 mg if ≥50 kg or 15 mg if <50 kg per manufacturer dosing) or IV placebo (saline). If assigned to the study arm, IV ketorolac will be administered by the anesthesia provider. All enrolled patients will receive standard post-operative pain management. Patients will be contacted post-operatively, to access pain scores and record the amount of the prescribed narcotic medications utilized since discharge.
  Interventions: Drug: Ketorolac (Toradol)
- Standard post-operative pain management + Placebo (saline) (Placebo Comparator): Subject will undergo an IVF cycle with ovarian hyperstimulation and oocyte retrieval. Standard protocols will be used for both study groups and involve administration of gonadotropins to stimulate ovarian follicle growth and regular monitoring with ultrasound and serum estradiol and progesterone levels until follicles reach a desired size. HCG or leuprolide acetate will be administered to trigger final oocyte maturation prior to oocyte retrieval under anesthesia. On the day of oocyte retrieval, the anesthesia provider will provide syringes of IV ketorolac (30 mg if ≥50 kg or 15 mg if <50 kg per manufacturer dosing) or IV placebo (saline). If assigned to the control arm, IV placebo (saline) will be administered by the anesthesia provider. All enrolled patients will receive standard post-operative pain management. Patients will be contacted post-operatively, to access pain scores and record the amount of the prescribed narcotic medications utilized since discharge.
  Interventions: Other: Placebo (saline)

INTERVENTIONS:
Drug: Ketorolac (Toradol) — IV Ketorolac (Toradol) will be administered at conclusion of oocyte retrieval. All enrolled patients will receive standard post-operative pain management.
  Arms: Standard post-operative pain management + Ketorolac (Toradol)
Other: Placebo (saline) — IV Placebo (saline) will be administered at conclusion of oocyte retrieval. All enrolled patients will receive standard post-operative pain management.
  Arms: Standard post-operative pain management + Placebo (saline)

SUMMARY:
To determine if a nonsteroidal anti-inflammatory drug (NSAID), Ketorolac (Toradol), can improve pain control and decrease narcotic use after undergoing egg retrieval.

DETAILED DESCRIPTION:
Postoperative pain control is an essential component to any surgical procedure. Surgery represents a time during which opioid-naïve patients may be exposed to narcotics, risking opioid related complications and future opioid-use disorder. Approximately 150,000 oocyte retrievals are performed per year in the United States, according to the 2017 Assisted Reproductive Technology National Summary Report. A reduction in exposure to narcotics in this field has significant public health implications, particularly given that approximately 6% of new persistent opioid use occurs following minor surgical procedures.

Ketorolac (Toradol) has been demonstrated to be a safe and efficacious agent to achieve pain control postoperatively with no significant increase in adverse events.

The purpose of this prospective randomized blinded placebo controlled trial is to determine if a nonsteroidal anti-inflammatory drug (NSAID), Ketorolac (Toradol), can improve pain control and decrease narcotic use after undergoing egg retrieval.

Approximately 400 women (n=200 in each arm) will be enrolled according to the inclusion/exclusion criteria among patients of Shady Grove Fertility. Participants will undergo a standard in vitro fertilization cycle (IVF) followed by egg retrieval (ER). Participants will be randomized to receive either IV ketorolac or IV placebo at the conclusion of the egg retrieval, administered by the anesthesia provider. All enrolled patients will receive standard post-operative pain management. The investigational component of this study lies in assessing post-operative pain control in the immediate post-operative period and in the post-operative period after discharge as reflected by pain scores and narcotic medication usage.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Females over 18 years of age who are scheduled to undergo oocyte retrieval
3. Patients must be able to read and understand written English or have an appropriate certified medical translator available.
4. Standard eligibility criteria to undergo IVF and embryo transfer at Shady Grove

Exclusion Criteria:

1. Known allergy to ketorolac
2. Those with known medical conditions precluding them from ketorolac use (active peptic ulcer disease, recent or history of hemorrhage or perforation, known renal or hepatic insufficiency, suspected or confirmed cerebrovascular bleeding, hemorrhagic diathesis, bleeding disorders, recent myocardial infarction, or stroke.)
3. BMI ≥ 40 kg/m2
4. History of substance abuse
5. Chronic opioid use
6. Transabdominal oocyte retrieval

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only female subjects will be recruited for this study as an oocyte retrieval requires ovary(ies) to be present and therefore this is only possible in the biological female sex.
Enrollment: 400 (Estimated)
Dates: Start 2022-08-10 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Administration of IV narcotic for rescue analgesia during recovery in the post anesthesia care unit (PACU) | Oocyte retrieval procedure day
  The primary objective is to evaluate the use of ketorolac as a safe and effective analgesic after transvaginal oocyte retrieval (TVOR) by assessing the number of patients requiring additional analgesia with IV narcotic during recovery in the post anesthesia care unit (PACU).

SECONDARY OUTCOMES:
Dose of narcotic for rescue analgesia during recovery in the PACU | Oocyte retrieval procedure day
  Dose of narcotic administered for rescue analgesia during recovery in the PACU
Type of narcotic for rescue analgesia during recovery in the PACU | Oocyte retrieval procedure day
  Type of narcotic administered for rescue analgesia during recovery in the PACU
Intensity of pain at baseline | Oocyte retrieval procedure day
  Pain (measured on a scale of 0 (no pain) to 10 (worst pain imaginable)): baseline pain score
Intensity of pain in PACU | Oocyte retrieval procedure day
  Pain (measured on a scale of 0 (no pain) to 10 (worst pain imaginable)): PACU pain scores (scored 0-10)
Intensity of pain after discharge | From oocyte retrieval procedure day up to 1 week post oocyte retrieval
  Pain (measured on a scale of 0 (no pain) to 10 (worst pain imaginable)): Home pain scores (scored 0-10)
Home narcotic use | From oocyte retrieval procedure day up to 1 week post oocyte retrieval
  Home post-operative narcotic use (recorded as number of pills)
Incidence of complications and adverse events | From oocyte retrieval procedure day up to 1 week post oocyte retrieval
  Data will be collected on the oocyte retrieval procedure including complications and adverse events in the intra-operative and post-operative periods
Biochemical pregnancy rate for patients who proceed to a fresh embryo transfer. | From date of randomization until ~10 days following embryo transfer
  Biochemical pregnancy is defined as the detection of beta HCG above 5 IU/L
Clinical pregnancy rate for patients who proceed to a fresh embryo transfer. | From date of randomization until 5-8 weeks estimated gestational age
  Clinical pregnancy is defined as the presence of a gestational sac(s)
Implantation rate for patients who proceed to a fresh embryo transfer. | From date of randomization until 7-8 weeks estimated gestational age
  Implantation rate is defined as the maximum number of gestational sacs per patient
Ongoing implantation rate for patients who proceed to a fresh embryo transfer. | From date of randomization until 7-8 weeks estimated gestational age
  The ongoing implantation rate is defined as maximum number of fetal heartbeats divided by total number of embryos transferred
Pregnancy loss rate for patients who proceed to a fresh embryo transfer. | From date of randomization until pregnancy loss, assessed up to 11 months
  Miscarriage; either biochemical or clinical pregnancy loss. Biochemical pregnancy loss is defined as initial positive beta HCG that did not progress to clinical pregnancy. Clinical pregnancy loss is defined as clinical pregnancy not progressing to live birth. Total pregnancy loss is defined as biochemical and clinical pregnancy loss (initial positive beta HCG that did not progress to live birth).
Live birth rate for patients who proceed to a fresh embryo transfer. | From date of randomization until live born infant at an estimated gestational age of at least 23 weeks or greater, assessed up to 11 months
  Live birth is defined as birth of a liveborn infant at an estimated gestational age of at least 23 weeks or greater.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Devine, MD, Principal Investigator — Shady Grove Fertility Reproductive Science Center
Locations (2):
- United States (2):
  - Shady Grove Fertility Reproductive Science Center, Rockville, Maryland
  - Shady Grove Fertility Reproductive Science Center, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waljee JF, Li L, Brummett CM, Englesbe MJ. Iatrogenic Opioid Dependence in the United States: Are Surgeons the Gatekeepers? Ann Surg. 2017 Apr;265(4):728-730. doi: 10.1097/SLA.0000000000001904. No abstract available. PMID 27429023
- [Background] Centers for Disease Control and Prevention. 2017 Assisted Reproductive Technology National Summary Report. US Dept of Health and Human Services; 2021.
- [Background] Wilson N, Kariisa M, Seth P, Smith H 4th, Davis NL. Drug and Opioid-Involved Overdose Deaths - United States, 2017-2018. MMWR Morb Mortal Wkly Rep. 2020 Mar 20;69(11):290-297. doi: 10.15585/mmwr.mm6911a4. PMID 32191688
- [Background] Kiani Z, Simbar M, Hajian S, Zayeri F. The prevalence of depression symptoms among infertile women: a systematic review and meta-analysis. Fertil Res Pract. 2021 Mar 4;7(1):6. doi: 10.1186/s40738-021-00098-3. PMID 33663615
- [Background] Kato T, Sampei M, Saito K, Morisaki N, Urayama KY. Depressive symptoms, anxiety, and quality of life of Japanese women at initiation of ART treatment. Sci Rep. 2021 Apr 6;11(1):7538. doi: 10.1038/s41598-021-87057-6. PMID 33824373
- [Background] Walter JR. Ketorolac use after oocyte retrieval: doing our part to combat the opioid crisis. F S Rep. 2021 Mar 12;2(2):142-143. doi: 10.1016/j.xfre.2021.03.001. eCollection 2021 Jun. No abstract available. PMID 34278342
- [Background] Brown CR, Moodie JE, Wild VM, Bynum LJ. Comparison of intravenous ketorolac tromethamine and morphine sulfate in the treatment of postoperative pain. Pharmacotherapy. 1990;10(6 ( Pt 2)):116S-121S. PMID 2082307
- [Background] Gobble RM, Hoang HLT, Kachniarz B, Orgill DP. Ketorolac does not increase perioperative bleeding: a meta-analysis of randomized controlled trials. Plast Reconstr Surg. 2014 Mar;133(3):741-755. doi: 10.1097/01.prs.0000438459.60474.b5. PMID 24572864
- [Background] Greer IA. Effects of ketorolac tromethamine on hemostasis. Pharmacotherapy. 1990;10(6 ( Pt 2)):71S-76S. PMID 2082316
- [Background] Maslin B, Lipana L, Roth B, Kodumudi G, Vadivelu N. Safety Considerations in the Use of Ketorolac for Postoperative Pain. Curr Drug Saf. 2017;12(1):67-73. doi: 10.2174/1574886311666160719154420. PMID 27440142
- [Background] Kang J, Chapdelaine P, Laberge PY, Fortier MA. Functional characterization of prostaglandin transporter and terminal prostaglandin synthases during decidualization of human endometrial stromal cells. Hum Reprod. 2006 Mar;21(3):592-9. doi: 10.1093/humrep/dei400. Epub 2005 Dec 8. PMID 16339169
- [Background] Mesen TB, Kacemi-Bourhim L, Marshburn PB, Usadi RS, Matthews M, Norton HJ, Hurst BS. The effect of ketorolac on pregnancy rates when used immediately after oocyte retrieval. Fertil Steril. 2013 Sep;100(3):725-8. doi: 10.1016/j.fertnstert.2013.04.048. Epub 2013 May 28. PMID 23721715
- [Background] Seidler EA, Vaughan DA, Leung AQ, Sakkas D, Ryley DA, Penzias AS. Routine ketorolac at oocyte retrieval decreases postoperative narcotic use by more than 50. F S Rep. 2021 Feb 10;2(2):156-160. doi: 10.1016/j.xfre.2021.02.003. eCollection 2021 Jun. PMID 34278347
- [Background] Siristatidis CS, Basios G, Pergialiotis V, Vogiatzi P. Aspirin for in vitro fertilisation. Cochrane Database Syst Rev. 2016 Nov 3;11(11):CD004832. doi: 10.1002/14651858.CD004832.pub4. PMID 27807847